CLINICAL TRIAL: NCT02191345
Title: A Randomized Controlled Trial Measuring the Effectiveness of Prerecorded Guided Imagery in Reducing Compassion Fatigue, Burnout, Perceived Stress, and State Anxiety of a Mental Health Nonprofit's Employees
Brief Title: The Effectiveness of Guided Imagery for a Nonprofit's Employees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FrontLine Service (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kimberly Juhas, Community Research Scholar, FrontLine Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MD002265; IRB-2014-743 (Other: Case Western Reserve University IRB)
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Focus of Study; Stress
Keywords: guided imagery; burnout; compassion fatigue; state anxiety
MeSH Terms: conditions — Burnout, Psychological; Compassion Fatigue; Anxiety Disorders | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10 minute break (No Intervention): Participants asked to take a 10 minute break as usual 3 times per week for 4 weeks
- Guided Imagery (Experimental): Participants listen to one of 6 pre-recorded guided imagery tracks 3 times per week for 4 weeks
  Interventions: Behavioral: Guided Imagery

INTERVENTIONS:
Behavioral: Guided Imagery — Guided imagery is a stress management technique that uses verbal suggestion and descriptive language to guide the listener into imagining sensations and visualizing images in the mind in order to bring about a desired physical response, such as reduction in anxiety, stress, or pain. The guided imagery tracks chosen for the study were chosen because their goal is relaxation and stress relief, and their length is under 15 minutes.
  Arms: Guided Imagery

SUMMARY:
Primary Aim A. To determine if listening to prerecorded guided imagery 3 times per week for 4 weeks will reduce state anxiety, perceived stress, burnout, compassion fatigue, and vicarious trauma in Fronltine Service staff.

Primary Aim B. To determine if staff will continue to listen to guided imagery after the first 4 weeks of the study is over.

DETAILED DESCRIPTION:
The purpose of this study is to compare the change in stress levels of employees who listen to prerecorded guided imagery to employees who take breaks, and to determine if employees are likely to adopt prerecorded guided imagery as a self-care tool.

Participants will be randomly assigned to either the guided imagery group or the control group. Members of the control group will be asked to take a 10 minute break 3 times per week for 4 weeks. Members of the guided imagery group will be asked to listen to one prerecorded guided imagery track 3 times per week for 4 weeks. All participants will fill out questionnaires before and after the 4 week period. All participants will fill out a short form before and after listening to each guided imagery, or before and after taking each break.

Phase 2: After phase 1 is complete, all participants will have the option to participate in phase 2 of the study. During phase 2, participants will receive a calendar and put a mark on every day that they listen to a guided imagery track. At the end of 4 weeks, participants will turn in the calendar.

ELIGIBILITY:
Inclusion Criteria:

* Staff of a nonprofit who work a minimum of three shifts per week
* Willing and able to use about 8-15 minutes of their lunch hours three times per week for for four weeks for the study

Exclusion Criteria:

* Staff members will be excluded from the study if they currently listen to guided imagery
* Those currently experiencing drug or alcohol abuse, suicidal ideation, or other serious mental health issue while not under the care of a trained mental health professional will also be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
State Anxiety as Measured by the State Anxiety Short Form | 4 weeks
  Participants in the experimental group will fill out the State Anxiety Short Form, a 6-item questionnaire before and after listening to guided imagery. Participants in the control group will fill out the same measure before and after taking a break.
  This will be done 3 times per week for a duration of 4 weeks.

SECONDARY OUTCOMES:
Compassion Fatigue, Compassion Satisfaction, and Burnout, as measured by the ProQol | 4 weeks
  Participants in both the control and experimental groups will complete the ProQol, a 30-item questionnaire, before and after the 4-week intervention period.
Perceived Stress as measured by the Perceived Stress Scale | 4 weeks
  Participants in the experimental and control groups will complete the Perceived Stress Scale, a self-report, 10-item questionnaire, before and after the 4-week intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Ashwini Sehgal, MD, Study Director — Case Western Reserve University, MetroHealth Medical Center; Kimberly A Juhas, MA, Principal Investigator — FrontLine Service
Locations (1):
- FrontLine Service, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No